CLINICAL TRIAL: NCT02159820
Title: Addition of Decitabine to Carboplatin-Paclitaxel in First-Line Treatment of Advanced Ovarian Cancer: A Phase 2-3, Open-label, Randomised Controlled Trial
Brief Title: Lower Dose Decitabine (DAC)-Primed TC (Carboplatin-Paclitaxel) Regimen in Ovary Cancer
Acronym: DAC and CT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, professor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PLA-BT-010; PLA-S-062
Record Dates: First submitted 2014-06-01; First posted 2014-06-10 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Primary Malignant Neoplasm of Ovary; FIGO Stages II to IV
MeSH Terms: interventions — Decitabine; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DTC Arm (Active Comparator): Patients are randomly assigned to receive lower-dose decitabine treatment followed by TC regimen (ie, DTC arm).
  Interventions: Drug: Decitabine (DTC Arm)
- TC regimen (Active Comparator): Patients were randomly assigned to receive carboplatin plus paclitaxel (ie, TC arm).
  Interventions: Drug: Paclitaxel and Carboplatin (TC Arm)

INTERVENTIONS:
Drug: Decitabine (DTC Arm) — Patients in DTC arm will receive lower-dose decitabine (7 mg/m2) administered intravenously within 1 hour for a consecutive 5 days, followed by TC regimen on day 6.
  Arms: DTC Arm
Drug: Paclitaxel and Carboplatin (TC Arm) — The TC arm consisted of paclitaxel 150 mg/m2 administered intravenously (IV) over 3 hours followed by carboplatin (area under the curve [AUC] 5) administered by IV over 30 to 60 minutes both on day 1 of a 3-week schedule. Dose reductions were allowed depending on hematologic or nonhematologic toxicity, as follows: carboplatin AUC4; paclitaxel 135 mg/m2. Patients who achieved partial remission after six cycles could receive additional cycles on their physicians' discretion.
  Arms: TC regimen

SUMMARY:
Ovarian cancer is the most lethal gynecological cancer and the 5th leading cause of cancer death in women. Most patients are typically diagnosed with advanced-stage disease. Platinum-paclitaxel regimen has been widely adopted as a standard first-line treatment for advanced ovarian cancer. Multiple collaborative randomised phase III trials evaluating the addition of a third chemotherapy agent, maintenance therapy or alternative taxanes failed to demonstrate significant improvements over a standard carboplatin/taxane doublet.

Decitabine (DAC), one major DNA demethylating agent, has been approved for treatment of preleukemic hematological disease myelodysplastic syndrome (MDS) by the Food and Drug Administration. Past trials of these with high doses, i.e., the use of maximal tolerated dose, for patients with solid tumors showed a low therapeutic index, due to extreme toxicities that have probably confounded the ability to document the true clinical response.

Low dose DNA demethylation agent decitabine (DAC) can resensitize the therapeutic indexes of resistent ovary cancer cells in vivo and in vitro.

The investigators hypothesized that DAC-triggered epigenetic reprogramming of tumor cells and possible immune cells could induce pronounced long-dated clinical effect by chemosensitization- and immunopotentiation-driven maximal eradicating roles on the minimal/residual lesions in primary patients with poor prognosis.

DETAILED DESCRIPTION:
Given the poor prognosis and the currently existed therapeutic strategies, The investigators will perform a prospective, randomized, phase II to III, intergroup trial to compare carboplatin plus paclitaxel (TC) with the DAC-primed TC (DTC) regimen in previously untreated patients with stage II to IV ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed International Federation of Gynecology and Obstetrics (FIGO) stages II to IV fallopian tube cancer, or primary peritoneal cancer. If only the results of cytological examinations were available, patients needed to have the following criteria: a cytological diagnosis of adenocarcinoma; an abdominal mass more than 2 cm in diameter on abdominal images; and a CA125 to carcinoembryonic antigen (CEA) ratio10 of more than 25, or no evidence of gastrointestinal cancer if CA125/CEA ratio was less than or equal to 25. Previous chemotherapy was not allowed.
* All patients had to be at least 18 years of age, to have an Eastern Cooperative
* Oncology Group (ECOG) performance status of 0-3, and were required to have adequate hematologic, renal, and hepatic function.

Exclusion Criteria:

* Patients were excluded if they had an ovarian tumour with a low malignant potential, or synchronous or metachronous (within 5 years) malignant disease other than carcinoma in situ.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2014-06; Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival in DTC treated advanced ovary cancer | up to 20 months
  The primary endpoint of this trial was progression-free survival (PFS), defined as the time from the date of randomisation to the date of the first occurrence of any of the following events: appearance of any new lesions that could be measured or assessed clinically; or CA125 criteria of disease progression. For patients with measurable disease, clinical or radiographical tumour measurements had priority over CA125 levels, and progression during treatment could not be declared on the basis of CA125 alone.
Overall survival rate in DTC treated advanced ovary cancer | 30 months
  Overall survival (OS), defined as the time from random assignment to death as a result of any cause, response rate, and adverse events.response to treatment, toxicity, and quality of life. Toxicities were evaluated per course and per patient (worst score over all courses).
Overall response rate in DTC treated advanced ovary cancer | 1 year
  Tumor measurements were made before each cycle by physical examination, before every third cycle by imaging methods in patients with measurable or evaluable disease, and after the last cycle. The same tumor assessment methods that were employed for baseline measurement were used for each repeat evaluation. Tumor response was graded according to Response Evaluation Criteria in Solid Tumors (RECIST).
Toxicity in DTC treated advanced ovary cancer | 8 months
  Adverse events and toxicities were graded according to the National Cancer Institute Common Toxicity Criteria (NIC-CTC). Toxicities were recorded continuously; blood chemistry parameters were measured before each treatment cycle and weekly thereafter.Quality of life was assessed with the use of the European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 and QLQ-OV28 questionnaires.

SECONDARY OUTCOMES:
Pharmacokinetics of lower-dose decitabine | up to 8 weeks
  Blood samples were obtained prior to treatment and at 0.25, 0.5, 1, 2, 4, 6, 8, and 24 hours after the first and fifth dose of decitabine. Plasma samples were stored and processed and further analyzed utilizing liquid chromatography/tandem mass spectrometry.
  Peak plasma concentration (Cmax) or area under the plasma concentration versus time curve (AUC) will be obtained from more than 10 patients treated at a decitabine dose level of 7mg/m2/d.

OTHER OUTCOMES:
Pharmacodynamics of lower-dose decitabine | up to 8 weeks
  To assess the pharmacodynamics of decitabine and to establish its relationship to clinical PFS, before and after decitabine treatment, peripheral blood mononuclear cells and/or tumor samples will be harvested for measurement of the expression and methylation profile including genes such as MLH1, RASSF1A, HOXA10, and HOXA11 by quantitative polymerase chain reaction (qPCR) and methylation-sensitive PCR analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Yuanguang Meng, Professor, Principal Investigator — Chinese PLA General Hospital; Weidong Han, professor, Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Fan H, Lu X, Wang X, Liu Y, Guo B, Zhang Y, Zhang W, Nie J, Feng K, Chen M, Zhang Y, Wang Y, Shi F, Fu X, Zhu H, Han W. Low-dose decitabine-based chemoimmunotherapy for patients with refractory advanced solid tumors: a phase I/II report. J Immunol Res. 2014;2014:371087. doi: 10.1155/2014/371087. Epub 2014 May 21. PMID 24963497
- See also: to recruit patients and let more oncologists know this trial — http://www.cancer.gov